CLINICAL TRIAL: NCT03097523
Title: Validation of a Cephalad Fluid Shift Countermeasure: Selection of Optimal Thigh Cuff Design Followed by Intracranial Pressure (ICP) Measurements During Extended Thigh Cuff Application
Brief Title: Mitigating Cephalad Fluid Shifts: A NSBRI Study
Acronym: NSBRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint John's Cancer Institute (Other)
Collaborators: National Space Biomedical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JWCI-16-0501
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Intracranial Pressure
Keywords: NSBRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Patients with intraventricular catheter meeting eligibility criteria will undergo the following procedures:
  * Blood pressure, heart rate, electrocardiogram and Intracranial Pressure (ICP) monitoring after standard of care procedures are completed
  * Continuous ICP monitoring using a disposable pressure transducer (i.e., TruWaveTM)
  * Sequential placement in an upright, seated, supine 0°, and supine 15° head down tilt (HDT) positions for approximately 15 minutes for stabilization, followed by: Non-invasive ICP, intra-ocular pressure (IOP) assessment, femoral vascular ultrasound, jugular vascular ultrasound, and assessment of adverse events
  Interventions: Device: Custom Thigh Cuff

INTERVENTIONS:
Device: Custom Thigh Cuff — The aim is to achieve positive and near normal forward arterial vascular blood flow to the lower extremities. Milder cuff pressures up to 65 mmHg will be used to limit venous return to the upper body.

SUMMARY:
This is a feasibility study to determine optimal thigh cuff design using a cephalad fluid shift protocol in patients who have an intraventricular catheter (such as Ommaya reservoir) placed for the delivery of central nervous system chemotherapy or for diagnosing potential elevation of ICP and monitoring its progression as part of standard medical care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-89 years old
* Willing and able to provide informed consent
* Patients who have an intraventricular catheter placed for the delivery of central nervous system chemotherapy or for diagnosing potential elevation of ICP and monitoring its progression as part of standard medical care
* KPS ≥ 70
* For patients on active anti-cancer (intra-thecal or IV) therapy, must be at least 2 weeks since last treatment; oral therapy is permitted

Exclusion Criteria:

* Less than 2 weeks since any prior surgery
* ICP > 20 mmHg that cannot be clinically stabilized
* Pregnant (Note: women of child-bearing potential must have a negative urine pregnancy test; women who are not of child-bearing potential are defined as: post-menopausal, age > 55 years with cessation of menses for 12 or more months; or less than 55 years with postmenopausal status confirmed by follicle-stimulating hormone in the post-menopausal range; or who have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy)
* Existing cardiovascular disease, diabetes, syncope, ocular disease that, in the opinion of the investigator, may confound the study results
* Uncontrolled neurological symptoms such as headache, nausea or vomiting that, in the opinion of the investigator, will limit the patient's ability to participate in the study
* Injury, trauma, venous thromboembolism, peripheral arterial disease or any condition that, in the opinion of the investigator, will prevent the subject from tolerating the application of a thigh cuff; history of treated DVT is permitted

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in intracranial pressure using cerebral and cochlear fluid pressure (CCFP) analyser and a disposable pressure transducer | 20 minutes
  Noninvasive and invasive ICP monitoring following standard of care procedures requiring access to ventricular catheter

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD, PhD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- John Wayne Cancer Institute at Providence Saint John's Health Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No
Data transfers or sharing is restricted to those JWCI study personnel identified on the site delegation log and/or per data use agreements. Data will be provided to the study sponsor.